CLINICAL TRIAL: NCT04794842
Title: Comparing Topical Tetracaine Drops to Topical Focal Phenol for Local Anesthesia During Intratympanic Steroid Injection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center - New Orleans (Unknown)
Responsible Party: Principal Investigator, Leslie Son, Academic Research Director, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tetracaine_vs_Phenol
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Intratympanic Steroid Injection; Idiopathic Sudden Sensorineural Hearing Loss; Meniere Disease
MeSH Terms: conditions — Meniere Disease | interventions — Tetracaine; Phenol

STUDY DESIGN:
Intervention Model Description: Single-Blinded Randomized Cohort
Who Masked: Participant
Masking Description: Intervention choice blinded to the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tetracaine (Active Comparator): Patients will be positioned in supine position at this time 0.5% tetracaine drops will be used to fill the ear canal. Tetracaine will then be allowed to stay in place for approximately 10 to 15 minutes with the patient's head positioned with affected ear up. After this, using an operative microscope the drops will be removed from the ear canal with suction.
  Interventions: Drug: Tetracaine 5% drops
- Phenol (Active Comparator): Patients will be positioned in supine position and tympanic membrane visualized with operative microscope. Phenol applicator will be used to topically apply 90% phenol to the injection site (posterior/Inferior aspect of tympanic membrane).
  Interventions: Drug: Phenol 90% concentration

INTERVENTIONS:
Drug: Tetracaine 5% drops — same as information in the arm/group description
  Arms: Tetracaine
Drug: Phenol 90% concentration — same as information in the arm/group description
  Arms: Phenol

SUMMARY:
Intratympanic steroid injections are an accepted treatment for Meniere's disease and idiopathic sudden sensorineural hearing loss. This treatment is typically performed using local topical anesthesia. There is very limited research on the differences of medications and application procedures effect on patients' pain during the procedure.Topical Tetracaine solution and topical phenol have been shown to be effective as local anesthesia for the tympanic membrane when used for myringotomy. Currently there is no consensus on medication and technique however focally applied phenol is the more widely used technique. We believe this study can provide valuable information given the disadvantages of topical phenol including burning upon application as well as possible increase in persistent tympanic membrane perforation. The objectives are to determine the effectiveness of tetracaine drops for local anesthesia for intratympanic steroid injections compared to focal topical phenol application and to identify if tetracaine drops provides adequate anesthesia for intratympanic steroid injection with less pain on application than focal phenol.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years of age or greater)
* Diagnosed with Idiopathic Sudden Sensorineural hearing loss or Meniere's disease
* Care plan includes treatment via intratympanic steroid injection

Exclusion Criteria:

* Having a current tympanic membrane perforation
* Adults unable to sign written consent
* Individuals less than 18 years of age
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Pain Score | Immediately following the procedure to 6 months from procedure
  Evaluate any differences in pain scores assessed pre/post intervention and between the two topical anesthetics used prior to the intratympanic steroid injection

SECONDARY OUTCOMES:
Statistical difference in tympanic membrane perforation presence or absence after the steroid injection procedure when using either tetracaine or phenol as the local anesthetic | Immediately following the procedure to 6 months from procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady of the Lake Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filipo R, Attanasio G, Russo FY, Viccaro M, Mancini P, Covelli E. Intratympanic steroid therapy in moderate sudden hearing loss: a randomized, triple-blind, placebo-controlled trial. Laryngoscope. 2013 Mar;123(3):774-8. doi: 10.1002/lary.23678. Epub 2013 Feb 1. PMID 23378346
- [Background] Wu HP, Chou YF, Yu SH, Wang CP, Hsu CJ, Chen PR. Intratympanic steroid injections as a salvage treatment for sudden sensorineural hearing loss: a randomized, double-blind, placebo-controlled study. Otol Neurotol. 2011 Jul;32(5):774-9. doi: 10.1097/MAO.0b013e31821fbdd1. PMID 21646929
- [Background] Leng Y, Liu B, Zhou R, Liu J, Liu D, Zhang SL, Kong WJ. Repeated courses of intratympanic dexamethasone injection are effective for intractable Meniere's disease. Acta Otolaryngol. 2017 Feb;137(2):154-160. doi: 10.1080/00016489.2016.1224920. Epub 2016 Sep 21. PMID 27650470
- [Background] McRackan TR, Best J, Pearce EC, Bennett ML, Dietrich M, Wanna GB, Haynes DS, Labadie RF. Intratympanic dexamethasone as a symptomatic treatment for Meniere's disease. Otol Neurotol. 2014 Oct;35(9):1638-40. doi: 10.1097/MAO.0000000000000500. PMID 25188506
- [Background] Belhassen S, Saliba I. Pain assessment of the intratympanic injections: a prospective comparative study. Eur Arch Otorhinolaryngol. 2012 Dec;269(12):2467-73. doi: 10.1007/s00405-011-1897-z. Epub 2011 Dec 28. PMID 22203120
- [Background] Silverstein H, Call DL. Tetracaine base. An effective surface anesthetic for the tympanic membrane. Arch Otolaryngol. 1969 Aug;90(2):150-1. doi: 10.1001/archotol.1969.00770030152010. No abstract available. PMID 5794873
- [Background] Kumar R, Banerjee A. Myringotomy and ventilation tube insertion with minims tetracaine drops. Eur Arch Otorhinolaryngol. 2011 Oct;268(10):1533-4. doi: 10.1007/s00405-011-1654-3. Epub 2011 Jun 17. PMID 21681571
- [Background] Hoffman RA, Li CL. Tetracaine topical anesthesia for myringotomy. Laryngoscope. 2001 Sep;111(9):1636-8. doi: 10.1097/00005537-200109000-00027. PMID 11568619
- [Background] Robertson A, Whitwell R, Osborne J. Is phenol a safe local anaesthetic for grommet insertion? J Laryngol Otol. 2006 Jan;120(1):20-3. doi: 10.1017/S0022215105005840. PMID 16375777
- [Background] Weisskopf A. Phenol anesthesia for myringotomy. Laryngoscope. 1983 Jan;93(1):114. doi: 10.1288/00005537-198301000-00022. No abstract available. PMID 6823169
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748